CLINICAL TRIAL: NCT06720259
Title: A Randomised, Single-Blinded Phase II Trial to Assess the Efficacy, Safety and Acceptability of Oxantel Pamoate in Comparison to Mebendazole for Trichuris Trichiura Infections in Children Aged 2-12 Years
Brief Title: Efficacy and Safety of Oxantel Pamoate in Children Infected With Trichuris Trichiura
Acronym: OXA-TRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Prof. Dr., Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OXA-TRI_1
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Trichuris Trichiura; Infection; Hookworm Infection; Ascaris Lumbricoides Infection
MeSH Terms: conditions — Trichuriasis; Hookworm Infections | interventions — oxantel pamoate; Mebendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxantel Single Dose (Experimental): Treatment with oxantel pamoate (20 mg/kg), orally administered on day 0
  Interventions: Drug: Oxantel Pamoate
- Oxantel Multiple Dose (Experimental): Treatment with oxantel pamoate (20 mg/kg), orally administered on each of day 0, 1 and 2
  Interventions: Drug: Oxantel Pamoate
- Mebendazole Single Dose (Active Comparator): Mebendazole (500mg), orally administered on day 0
  Interventions: Drug: Mebendazole

INTERVENTIONS:
Drug: Oxantel Pamoate — Tablets containing 250 mg oxantel pamoate
  Arms: Oxantel Multiple Dose; Oxantel Single Dose
Drug: Mebendazole — Tablets containing 500 mg mebendazole
  Arms: Mebendazole Single Dose

SUMMARY:
This study aims to provide evidence on the efficacy, safety and acceptability of the new, chewable formulation of oxantel pamoate administered as a single dose or multiple doses, compared to mebendazole in children infected with T. trichiura. This study will involve children aged 2-12 years, since an infection with T. trichiura occurs often in children.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2 and 12 years.
* Written informed consent signed by parents/caregivers (signature or thumbprint) and, for children aged 6-12 years, written assent from the child.
* Agree to comply with study procedures, including provision of two stool samples at the baseline and at follow-up assessment 14-21 days after treatment, respectively.
* At least two out of four Kato-Katz thick smears positive for T. trichiura at baseline.
* Willing to be examined by a study physician prior to treatment.

Exclusion Criteria:

* Presence or signs of major systemic illness or abnormal physical findings at screening, e.g. severe anaemia (Hb level <80 g/L according to WHO) upon initial clinical assessment.
* Known allergy to study medication (i.e. oxantel pamoate, mebendazole or any of the excipients).
* Use of anthelminthic drugs within 4 weeks before or during study period.
* Being prescribed or taking concomitantly medication with known contraindication or drug interactions with the study medication.
* Actively participating in other clinical trials during the study.
* Pregnancy (female participants that report to have reached menarche

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Cure rate (CR) of oxantel pamoate single dose compared to mebendazole T. trichiura | 14-21 days after treatment
  CR will be calculated as the percentage of Trichuris trichiura egg-positive participants at baseline who become egg-negative after treatment.

SECONDARY OUTCOMES:
Egg reduction rate (ERR) of oxantel pamoate single dose compared to mebendazole against T. trichiura | 14-21 days after treatment
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric and arithmetic mean egg counts will be calculated for the two treatment arms before and after treatment to assess the corresponding ERRs.
Cure rate (CR) and egg reduction rate (ERR) of oxantel pamoate multiple doses compared to oxantel single dose against T. trichiura | 14-21 days after treatment
  CR and ERR will be calculated as described in primary outcome measure and the first listed secondary outcome measure, respectively.
Cure rate (CR) and egg reduction rate (ERR) of oxantel pamoate multiple doses compared to mebendazole against T. trichiura | 14-21 days after treatment
  CR and ERR will be calculated as described in primary outcome measure and the first listed secondary outcome measure, respectively.
Cure rates (CRs) and egg reduction rates (ERRs) of oxantel pamoate compared to mebendazole against Ascaris lumbricoides and hookworm infections in co-infected participants | 14-21 days after treatment
  CR and ERR will be calculated as described in primary outcome measure and the first listed secondary outcome measure, respectively.
Number of adverse events (AE) to assess safety and tolerability of oxantel pamoate administered as a single dose or as multiple doses, and compared with mebendazole | 3 hours, 24 hours (and 48 and 72h for the multiple dose treatment arm) and 14-21 days after treatment
  Participants will be monitored at the site for 3 hours following treatment for any acute AEs. Participants will be interviewed 3 hours after treatment, as well as 24 hours after every dose received, as well as 14-21days after the last treatment dose about the occurrence of AEs.
  AEs will be evaluated descriptively as the difference of proportion reported AEs before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Keiser, PhD, Study Chair — Swiss Tropical & Public Health Institute
Locations (1):
- Public Health Laboratory Ivo de Carneri, Chake Chake, Tanzania